CLINICAL TRIAL: NCT01287689
Title: An Open, Uncontrolled, Non-interventional Observational Cohort Outcome Study of Immunoglobulins in 3 Indications: Primary and Secondary Immunodeficiencies and Neurological Auto-immune Diseases
Brief Title: Assessment of Immunoglobulins (IgG) in a Long-term Non-interventional Study
Acronym: SIGNS
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: SIGNS
Record Dates: First submitted 2011-01-24; First posted 2011-02-01 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Primary Immunodeficiency (PID); Secondary Immunodeficiency (SID); Neurological Autoimmune Disease
Keywords: Non-interventional trial; immunodeficiency; outcome study, registry; long-term outcomes, drug utilization; effectiveness, treatment patterns; patient characteristics under real life conditions; factors for treatment success; long-term tolerability; quality of life
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Immunologic Deficiency Syndromes | interventions — Immunoglobulin G

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient treated with any IgG: Any marketed SC or IV IgG can be documented
  Interventions: Other: Immunoglobulin G (IgG)

INTERVENTIONS:
Other: Immunoglobulin G (IgG) — Not applicable. All interventions are at the discretion of the investigator. All marketed IgG formulations can be documented.

SUMMARY:
This non-interventional, epidemiological study assesses long-term outcomes in subjects receiving immunoglobulins (IgG) for any treatment purpose, irrespective of the regimen prescribed by the treating physician, under routine clinical conditions in Germany.

Long-term outcome data are collected on patient characteristics in the various indications, drug utilization of intravenous and subcutaneous IgG (e.g. treatment and dosing patterns), effectiveness (i.e. number of infections), tolerability, health related quality of life, and economic variables (number of hospitalizations, sick-leave days etc.) with the possibility to estimate direct costs.

DETAILED DESCRIPTION:
In view of the broad range of indications in immunodeficiency and immunomodulation, it is of interest to document the use of IgG under the conditions of everyday practice and to analyze the endpoints (outcomes). A prospective cohort study such as this is an important evidence source for such rare diseases as those mentioned above. The aim of this outcome study is to fill the gap of the lack of long-term data in these rare diseases treated with IgG.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender with primary, severe secondary immunodeficiency and recurrent infections or neurological autoimmune diseases
* Naïve to IgG, or pre-treated with IgG
* Subject or parent/legally authorized representative has provided written informed consent.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ambulatory or hospital-based patients (no age restriction)
Sampling Method: Non-Probability Sample
Enrollment: 685 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Immunoglobulin IgG dosage | up to 54 months
  Dosage of immunoglobulins (IgG); frequency of IgG administrations; days of treatment with IgG; duration of infusion of IgG.

SECONDARY OUTCOMES:
Infection rate | up to 54 months
  For immunodeficiencies (primary PID and secondary SID):
  frequency of infections; degree of severity of infections (SBIs); duration of antibiotic treatment; necessity of antibiotic treatment.
Neurological and muscular function (for neurological auto-immune diseases only) | up to 54 months
  Grip strength (dynamometer) Electrophysiology (EMG, ENG); Inflammatory Neuropathy Cause and Treatment (INCAT) disability score; EDSS, annual relapse rate; Myasthenia Score.
Duration of manifest auto-immune disease within the follow-up period(for neurological auto-immune diseases only). | up to 54 months
Health-related quality of life | up to 54 months
Pharmacoeconomic parameters | up to 54 months
  Number of sick-leave days Number of medical visits Days of hospitalisation due to infections or due to disability or loss of function Degree of disability

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Kirch, MD, PhD, Principal Investigator — Institute for Clinical Pharmacology, Medical Faculty, Technical University Dresden, Germany; David Pittrow, MD, PhD, Study Chair — Institute for Clinical Pharmacology, Medical Faculty, Technical University, Dresden, Germany; Michael Borte, MD, PhD, Study Director — Fachbereich Pädiatrische Rheumatologie, Immunologie und Infektiologie am Klinikum St. Georg gGmbH Leipzig, Akademisches Lehrkrankenhaus der Universität Leipzig, Germany; Ulrich Baumann, MD, PhD, Study Director — Klinik für Pädiatrische Pneumologie, Allergologie und Neonatologie, Medizinische Hochschule Hannover (MHH), Germany; Manfred Hensel, MD, PhD, Study Director — Mannheimer Onkologie Praxis, Mannheim, Germany; Dörte Huscher, Study Director — Epidemiologie, Rheumaforschungszentrum Berlin, Germany; Marcel Reiser, MD, PhD, Study Director — PIOH - Praxis Internistische Onkologie, Hämatologie, Köln, Germany; Martin Stangel, MD, PhD, Study Director — Klinik für Neurologie, Medizinische Hochschule Hannover (MHH), Germany; Ralph Gold, MD, PhD, Study Director — Klinik für Neurologie, St. Josef-Hospital, Klinikum der Ruhr-Universität Bochum, Germany; Claudia Sommer, MD, PhD, Study Director — Neurologische Klinik und Poliklinik, Universitätsklinik Würzburg, Germany
Locations (7):
- Germany (7):
  - Klinik für Neurologie, St. Josefs-Hospital der Ruhr-Univ., Bochum
  - Praxis für Hämatologie und Internistische Onkologie, Cologne
  - Institute for Clinical Pharmacology, Dresden
  - Klinik für Neurologie, Medizinische Hochschule, Hanover
  - Klinik für Pädiatrische Pneumologie, Allergologie und Neonatologie, Medizinische Hochschule (MHH)., Hanover
  - Fachbereich Pädiatrische Rheumatologie, Immunologie und Infektiologie am Klinikum St. Georg gGmbH Leipzig, Akademisches Lehrkrankenhaus der Universität, Leipzig
  - Mannheimer Onkologie-Praxis, Mannheim

REFERENCES:
- [Background] Kirch W, Gold R, Hensel M, Fasshauer M, Pittrow D, Huscher D, Reiser M, Stangel M, Baumann U, Borte M. [Assessment of immunoglobulins in a long-term non-interventional study (SIGNS Study). Rationale, design, and methods]. Med Klin (Munich). 2010 Sep;105(9):647-51. doi: 10.1007/s00063-010-1105-8. Epub 2010 Sep 28. German. PMID 20878302
- [Result] Borte M, Baumann U, Pittrow D, Hensel M, Fasshauer M, Huscher D, Reiser M, Stangel M, Gold R, Kirch W; Liste der aktuell beitragenden Zentren, sortiert nach Postleitzahlen (mindestens ein Patient zum 1.3.2012). [Immunoglobulins in PID, SID and neurological autoimmune disease]. Dtsch Med Wochenschr. 2012 Mar;137(13):675-80. doi: 10.1055/s-0032-1304844. Epub 2012 Mar 20. German. PMID 22434180
- [Result] Stangel M, Baumann U, Borte M, Fasshauer M, Hensel M, Huscher D, Kirch W, Pittrow D, Reiser M, Gold R. Treatment of neurological autoimmune diseases with immunoglobulins: first insights from the prospective SIGNS registry. J Clin Immunol. 2013 Jan;33 Suppl 1:S67-71. doi: 10.1007/s10875-012-9789-6. Epub 2012 Sep 14. PMID 22976553
- [Result] Stangel M, Gold R, Pittrow D, Baumann U, Borte M, Fasshauer M, Hensel M, Huscher D, Reiser M, Sommer C. Treatment of patients with multifocal motor neuropathy with immunoglobulins in clinical practice: the SIGNS registry. Ther Adv Neurol Disord. 2016 May;9(3):165-79. doi: 10.1177/1756285616629869. Epub 2016 Feb 16. PMID 27134672
- [Result] Reiser M, Borte M, Huscher D, Baumann U, Pittrow D, Sommer C, Stangel M, Fasshauer M, Gold R, Hensel M. Management of patients with malignancies and secondary immunodeficiencies treated with immunoglobulins in clinical practice: Long-term data of the SIGNS study. Eur J Haematol. 2017 Aug;99(2):169-177. doi: 10.1111/ejh.12900. Epub 2017 Jun 21. PMID 28467615